CLINICAL TRIAL: NCT04602039
Title: The Anti-inflammatory Effects of Dairy Colostrum Neovite™ as a Dietary Supplement for Humans
Brief Title: Colostrum and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, Richard Bracken, Assoicate Professor, Swansea University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRAS190222
Record Dates: First submitted 2017-08-24; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; colostrum
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This was a non-randomised control trial involving individuals split into 3 groups (healthy, prediabetes, type 2 diabetes) that all received colostrum for 28 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- People without Diabetes (Experimental): A 4 week supply of a commercial dairy colostrum supplement (Neovite™) given to each participant.
  Interventions: Dietary Supplement: Bovine Colostrum
- Participants with Pre-diabetes (Experimental): A 4 week supply of a commercial dairy colostrum supplement (Neovite™) given to each participant.
  Interventions: Dietary Supplement: Bovine Colostrum
- Participants with Type 2 diabetes (Experimental): A 4 week supply of a commercial dairy colostrum supplement (Neovite™) given to each participant.
  Interventions: Dietary Supplement: Bovine Colostrum

INTERVENTIONS:
Dietary Supplement: Bovine Colostrum — Bovine colostrum (Neovite)

SUMMARY:
Colostrum is the milk that is first produced by a mother after giving birth. It plays a key role in the normal early development of mammals by providing substances that are important for nutrition, immunological defence and healthy growth and development. Research has shown that the immunoglobulins, antimicrobial peptides and growth factors in dairy colostrum and early season milk from cows are nearly identical to human. After puberty our bodies begin the aging process, and gradually produce less immune and growth factors that resist disease and heal tissue. Colostrum is a natural source of these life-enhancing components. Research shows that colostrum supports immune function and can help use fat for fuel and optimise cellular reproduction. Colostrum is receiving an increasing amount of interest in the healthcare community because of the potential benefits it can offer to a variety of patient groups by boosting the body's immune response, encouraging growth and repair in the gut, stabilising gut microflora and supporting better nutritional absorption and muscle growth.

Diabetes is a chronic condition associated with significant morbidity and mortality predominantly from associated chronic diseases. Currently within the UK approximately 5% of NHS spend is in relation to type 2 diabetes alone. Within Wales, approximately £256 million is spent on the care of these patients. Estimates suggest that people with type 2 diabetes have the disease for approximately 10 years before diagnosis, during which complications become well established including dyslipidaemia and hypertension. Additionally, many of these people are overweight or obese before they develop diabetes. The prevalence of type 2 diabetes continues to increase despite recent advances in our understanding of the basic physiology of glucose control. There is a clear association between inflammation, insulin resistance and type 2 diabetes. We aim to target inflammation levels seen in those with impaired glucose homeostasis such as impaired fasting glucose (IFG) and impaired glucose tolerance (IGT), collectively called pre-diabetes.

DETAILED DESCRIPTION:
Colostrum is the milk that is first produced by a mother after giving birth. It plays a key role in the normal early development of mammals by providing substances that are important for nutrition, immunological defence and healthy growth and development. Research has shown that the immunoglobulins, antimicrobial peptides and growth factors in dairy colostrum and early season milk from cows are nearly identical to human. After puberty our bodies begin the aging process, and gradually produce less immune and growth factors that resist disease and heal tissue. Colostrum is a natural source of these life-enhancing components. Research shows that colostrum supports immune function and can help use fat for fuel and optimise cellular reproduction. Colostrum is receiving an increasing amount of interest in the healthcare community because of the potential benefits it can offer to a variety of patient groups by boosting the body's immune response, encouraging growth and repair in the gut, stabilising gut microflora and supporting better nutritional absorption and muscle growth.

Diabetes is a chronic condition associated with significant morbidity and mortality predominantly from associated chronic diseases. Currently within the UK approximately 5% of NHS spend is in relation to type 2 diabetes alone. Within Wales, approximately £256 million is spent on the care of these patients. Estimates suggest that people with type 2 diabetes have the disease for approximately 10 years before diagnosis, during which complications become well established including dyslipidaemia and hypertension. Additionally, many of these people are overweight or obese before they develop diabetes. The prevalence of type 2 diabetes continues to increase despite recent advances in our understanding of the basic physiology of glucose control. There is a clear association between inflammation, insulin resistance and type 2 diabetes. We aim to target inflammation levels seen in those with impaired glucose homeostasis such as impaired fasting glucose (IFG) and impaired glucose tolerance (IGT), collectively called pre-diabetes.

The focus of the work will be to investigate the effects of dairy colostrum as a food supplement on inflammatory processes and the potential role that it could play in the prevention of pre-diabetes developing into type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* both genders

  * age 18-65 years
  * no impaired glucose homeostasis (HbA1c <6.0% or <42mmol/mol) (Group 1)
  * impaired fasting glucose (IFG) or impaired glucose tolerance (ITG) (HbA1c 6.0-6.5% or 42-48mmol/mol) (Group 2)
  * type 2 diabetes (>6.5% or >48mmol/mol) (Group 3)

Exclusion Criteria:

* those who cannot give informed consent

  * those who are lactose intolerant
  * females who are pregnant or breastfeeding
  * those with type 1 diabetes
  * those with chronic kidney disease
  * those taking GLP-1 agonists or DPP-4 inhibitors (gliptins)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
This project aimed to examine changes in insulin resistance in participants using dairy colostrum as a food supplement | before and after 28 days supplementation
  insulin resistance (HOMA-IR)

SECONDARY OUTCOMES:
This project aimed to examine changes in inflammatory markers in participants using dairy colostrum as a food supplement | before and after 28 days supplementation
  to measure CRP
This project aimed to examine changes in inflammatory markers in participants using dairy colostrum as a food supplement | before and after 28 days supplementation
  to measure IL6
This project aimed to examine changes in inflammatory markers in participants using dairy colostrum as a food supplement | before and after 28 days supplementation
  to measure iFABP

IPD SHARING:
Plan to Share IPD: No